CLINICAL TRIAL: NCT00192140
Title: An Open-Label, Single-Arm Trial to Assess the Shedding, Immunogenicity, and Safety of FluMist Administered to Healthy Individuals 5-49 Years of Age
Brief Title: Trial to Assess the Shedding,Immunogenicity, and Safety of FluMist Administered to Healthy Individuals 5-49 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Chris Ambrose, Dir. Medical Affairs, MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM026
Record Dates: First submitted 2005-09-09; First posted 2005-09-19 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): FluMist
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — A single intranasal dose of FluMist will be administered to approx. 300 subjects.

SUMMARY:
* To describe the proportion of individuals 5-49 years of age who shed vaccine strain viruses.
* To describe the duration of shedding of vaccine viruses in individuals 5-49 years of age.
* To describe the genotypic and phenotypic stability of shed vaccine viruses.
* To describe the immune responses of FluMist in individuals 5-49 years of age.
* To describe the safety of FluMist in individuals 5-49 years of age in relation to shedding and the immune response

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the viral shedding, immunogenicity and safety of FluMist when administered to healthy individuals between 5-49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 5-49 years of age;
* In good health;
* Individual or parent/guardian available by telephone;
* Ability of the participant or parent/guardian to understand and comply with the requirements of the protocol; and
* Signed informed consent and HIPAA authorization by the participant or parent/guardian.

Exclusion Criteria:

* History of hypersensitivity to any component of FluMist, including egg or egg products;
* History of hypersensitivity to gentamicin;
* Close contact who is immunocompromised within the same household;
* Known or suspected immune deficiency diseases or immunosuppressed or have altered or compromised immune status as a consequence of treatment with immunosuppressive therapies;
* History of chronic underlying medical conditions such as chronic disorders of the cardiovascular and pulmonary systems, chronic metabolic diseases (including diabetes), renal dysfunction, or hemoglobinopathies;
* History of Guillain-Barré syndrome;
* History of asthma or reactive airways disease;
* Acute febrile (>100.0°F oral) and/or respiratory illness, within the 72 hours prior to enrollment;
* For children and adolescents - use of aspirin or aspirin containing products in the month prior to enrollment or anticipated use during the study;
* Pregnancy or, in biologically capable women (e.g., menses within the last year), not willing to agree to acceptable birth control for three months after enrolling into the study (for those biologically capable, a urine pregnancy test must be performed on the day of vaccination with a negative result);
* Administration of any intranasal medication within two weeks prior to enrollment or expected receipt during this study;
* Administration of any live virus vaccine within one month prior to enrollment or if receipt of another live virus vaccine is expected within one month of the vaccination in this study;
* Administration of any inactivated vaccine within two weeks prior to enrollment or if receipt of another inactivated vaccine is expected within two weeks of the vaccination in this study;
* Participation in another investigational trial or administration of any investigational drug within one month prior to enrollment or during this study;
* Employees of the research center, any individuals involved with the conduct of the study, or any family member of such individuals;
* Laboratory confirmed influenza (positive culture or rapid antigen test) in the prior influenza season (2003/2004 or 2004/2005 season);
* Receipt of any influenza vaccine in the prior influenza season; and
* Any condition that in the opinion of the investigator would interfere with the interpretation or evaluation of the vaccine.

Ages: 5 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 345
Dates: Start 2004-06; Primary Completion 2004-10 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To describe the proportion of individuals 5-49 years of age who shed vaccine strain viruses. | 28 days after vaccination
To describe the duration of shedding of vaccine viruses in individuals 5-49 years of age. | 28 days after vaccination

SECONDARY OUTCOMES:
To describe the immune responses of FluMist in indivduals 5-49 years of age. | 28 days after vaccination
To describe the safety of FluMist in individuals 5-49 years of age in relation to shedding and the immune response. | 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — Sponsor GmbH
Locations (11):
- United States (11):
  - SFBC International, Inc, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Kentucky Pediatric / Adult Research, Inc, Bardstown, Kentucky
  - University of Maryland, School of Medicine, Baltimore, Maryland
  - Center for Vaccine Development, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Pediatric Clinical Trials International, Columbus, Ohio
  - Primary Physician's Research Inc., Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center North, Nashville, Tennessee
  - University of Virginia, Elson Student Health Center, Charlottesville, Virginia
  - Marshall University Medical Center, Huntington, West Virginia